CLINICAL TRIAL: NCT06825819
Title: DETERMINING THE IMPACT OF MICROBIAL DYSBIOSIS ON IMMUNE AND BARRIER DYSFUNCTION IN LONG COVID
Brief Title: Dysbiosis & Long COVID
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB24-1178
Record Dates: First submitted 2025-02-11; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects without Long COVID symptoms: We will enroll non-hospitalized patients recruited through the UCM long COVID clinic (headed by Dr. Rasika Karnik) and through the UCM Dept. of Gastroenterology endoscopy center under the umbrella Genesys protocol. We will also enroll convalescent subjects from the community without long COVID symptoms (only blood and stool samples collected from community participants, and they need not consent to the Genesys study to participate). All subjects will have had at least 1 PCR- or antigen-confirmed COVID-19 infection within the past 3 years and will be at least 60 days from their last SARS-CoV-2 infection.
  Interventions: Biological: Subjects with and without Long COVID
- Subjects with Long COVID symptoms: We will enroll non-hospitalized patients recruited through the UCM long COVID clinic (headed by Dr. Rasika Karnik) and through the UCM Dept. of Gastroenterology endoscopy center under the umbrella Genesys protocol. We will also enroll convalescent subjects from the community with long COVID symptoms (only blood and stool samples collected from community participants, and they need not consent to the Genesys study to participate). All subjects will have had at least 1 PCR- or antigen-confirmed COVID-19 infection within the past 3 years and will be at least 60 days from their last SARS-CoV-2 infection.
  Interventions: Biological: Subjects with and without Long COVID

INTERVENTIONS:
Biological: Subjects with and without Long COVID — To collect biospecimens (matched stool & blood) samples from 400 people with and without long COVID (200 participants/group) to understand how COVID-induced dysbiosis impacts symptom severity, immune suppression, and gut barrier dysfunction both ex vivo and in vitro.

SUMMARY:
The SARS-CoV-2 virus causes COVID-19, which ranges from mild initial symptoms to severe multi-organ dysfunction. While some patients recover to their baseline states, others develop a long COVID, or post-acute sequelae of SARS-CoV-2 (PASC) consisting of symptoms persisting >2-6 months post-infection. PASC symptoms include post-exertional malaise, fatigue, and heart palpitations as well as incident GI disorders, cognitive dysfunction, and arthritis. Based on prevalence/incidence studies, it is estimated that more than 30 million people in the US have ever developed PASC with 10-11% of patients or 11 million people continuing to feel symptoms to the present day10. SARS-CoV-2 vaccines are only ~32% effective against infection at 4 months post-vaccination11, only 15% effective against the development of PASC12, and only 20% of American adults have received an updated booster as of December 202313. It is therefore imperative that the scientific community make progress in identifying underlying causes of PASC to develop effective treatments.

This study will identify microbial metabolites associated with PASC-mediated gut dysbiosis and establish a tractable in vitro model to test T cell-gut epithelium dynamics to develop novel bio-therapeutics for multiple post-viral conditions. This case-control study will collect biospecimens (matched stool & blood) samples from 400 people with and without long COVID (200 participants/group) to understand how COVID-induced dysbiosis impacts symptom severity, immune suppression, and gut barrier dysfunction both ex vivo and in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80
* Sex: Any
* Race: Any
* Last COVID infection: within past 3 years, PCR- or antigen-confirmed, symptomatic (mild/moderate/severe)
* COVID vaccination status: Any
* Presence of long COVID symptoms (GI, cardiac, pulmonary, neuro, musculoskeletal, and/or psych): 200 with symptoms, 200 w/o symptoms as defined by SBQ-LCTM.
* May or may not be doing routine endoscopy at UCM

Exclusion Criteria:

* Age <18 or >80
* Last COVID infection >3 years ago (PCR/antigen-confirmed, symptomatic)
* Currently or within the last 3 months COVID+ by nasopharyngeal PCR/antigen test
* Currently diagnosed with cancer
* Currently pregnant (cannot take colon biopsy sample; only eligible for survey/blood & stool collection)
* Currently on biologic immunomodulatory medications
* Official diagnosis of irritable bowel disease (IBD) or other chronic GI disorder

Vulnerable and/or Special Populations

* Healthy adult volunteers
* Pregnant people
* UCMC and UChicago employees
* Staff/faculty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll non-hospitalized patients recruited through the UCM long COVID clinic (headed by Dr. Rasika Karnik) and through the UCM Dept. of Gastroenterology endoscopy center under the umbrella Genesys protocol. We will also enroll convalescent subjects from the community with and without long COVID symptoms (only blood and stool samples collected from community participants, and they need not consent to the Genesys study to participate). All subjects will have had at least 1 PCR- or antigen-confirmed COVID-19 infection within the past 3 years and will be at least 60 days from their last SARS-CoV-2 infection. We will recruit a total of 400 subjects (200 ea. w/ and w/o long COVID). The research will be conducted at UCM clinic sites and in laboratory facilities
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
To determine whether people with long COVID exhibit microbial dysbiosis characterized by decreased bacterial diversity, overgrowth of Bacteroides taxa, and lower SCFA, indole, and secondary bile acid production with biospecimen collections | At baseline until final values

SECONDARY OUTCOMES:
To collect matched stool, blood, and intestinal biopsy samples from a cohort of 300 individuals with and without long COVID (150/group) | At baseline until final values

OTHER OUTCOMES:
Viral persistence of SARS-CoV-2 in intestinal biopsies (RNAScope). | At baseline until final values
  This will only be done if participants consent to both this study and the Genesys study.
Composition of microbial taxa in stool (shotgun metagenomics) | At baseline until final values
Generation of colonic organoids; determination of barrier function +/- autologous metabolites, PBMCs, T cell stimulation, Spike pseudovirus infection (BSL-2). | At baseline until final values
  This will only be done if participants consent to both this study and the Genesys study.
Assessment of T cell metabolism by flow cytometry | At baseline until final values

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya Visvabharathy, Ph.D, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided